CLINICAL TRIAL: NCT06482866
Title: Risk Factors Leading to the Formation of Intranasal Synechiae in Patients After Endonasal Surgery
Brief Title: Synechie Afrer Rhinosug. Proc. 2024
Status: Completed | Type: Observational
Sponsor: Mateusz Jan Stępiński (Other)
Responsible Party: Sponsor-Investigator, Mateusz Jan Stępiński, Lek., Multidisciplinary Regional Hospital in Gorzow
Organization: Multidisciplinary Regional Hospital in Gorzow (Other)
Other Study IDs: SYNECHIE2024
Record Dates: First submitted 2024-06-26; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Complication of Surgical Procedure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Patients underwent septoconchoplasty with or without turbionplasty. Surgeons didn't use nasal splits.
  Interventions: Other: Cottle's septoplasty and radiocoagulation conchoplasty
- Study group: Patients underwent septoconchoplasty with or without turbionplasty. Surgeons used nasal splits.
  Interventions: Other: Cottle's septoplasty and radiocoagulation conchoplasty

INTERVENTIONS:
Other: Cottle's septoplasty and radiocoagulation conchoplasty — Cottle's septoplasty and radiocoagulation conchoplasty Study group - added nasal splits; Control group - nasal splits weren't used.

SUMMARY:
Analyze the factors influencing the development of intranasal adhesions (synechiae), with particular emphasis on the use of nasal septal separators, and to suggest a solution to reduce this complication in the future.

Analyze of the medical documentation. It was not an experimental examination.

ELIGIBILITY:
Inclusion Criteria:

* septo or septoconchoplasty

Exclusion Criteria:

* incompleted documentation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were operated in Polish hospital (Gorzów Wlkp).
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Synechie | Between 2 weeks to 12 month
  Intranasal synechiae after rhino nasal procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Multidisciplinary Regional Hospital, Gorzów Wielkopolski, Woj. Lubuskie, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Publication of results in open access magazine